CLINICAL TRIAL: NCT05929911
Title: Pilot Feasibility Proposal to Adapt Trauma-focused Psychodynamic Psychotherapy (TFPP) for PLWH and PTSD
Brief Title: Open Trial of Trauma-focused Psychodynamic Psychotherapy for People Living With HIV and PTSD
Acronym: TFPP-PLWH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); American Psychoanalytic Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-15016; P30AI124414 (NIH)
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder; HIV
Keywords: PTSD; HIV; psychotherapy; trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — 2,2,3,3-tetrafluoroputrescine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-focused psychodynamic psychotherapy (Experimental): Twice-weekly psychotherapy for 24 sessions
  Interventions: Behavioral: Trauma-focused psychodynamic psychotherapy

INTERVENTIONS:
Behavioral: Trauma-focused psychodynamic psychotherapy — This psychotherapy addresses disruptions in the ability to reflect and affective regulation by exploring the psychological meanings of symptoms and their relation to traumatic events. The therapist works to identify intrapsychic conflicts, intense negative affects, and defense mechanisms related to the PTSD syndrome using a psychodynamic formulation that provides a framework for intervention. The transference provides a forum for patients to address feelings of mistrust, difficulties with authority, fears of abuse, angry and guilty feelings, and fantasies.
  This treatment will be provided in-person or over teletherapy as the public health situation demands.
  Other Names: TFPP

SUMMARY:
People living with HIV (PLWH) have a higher rate of post-traumatic stress disorder (PTSD) diagnosis than the general population. Comorbid PTSD is also associated with negative HIV-related health outcomes. Unfortunately, little outcome research has examined the usefulness of PTSD treatments for PTSD. This pilot study adapts for PLWH a non-exposure based psychotherapy for PTSD focused on reflecting on one's emotions and relationships and understanding and working through how trauma may have disrupted them. The study team is interested in better understanding the needs of PLWH with PTSD, learning whether PLWH with PTSD find this treatment acceptable and helpful, and beginning to understand the relationship between HIV-related health factors (e.g., inflammation and stress biology) and PTSD, and how these health factors may improve during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DSM-5 defined PTSD, per the Clinician Administered PTSD Scale & CAPS-5 total severity score greater than or equal to 25
* HIV diagnosis (by medical records or HIV testing)
* Stable psychiatric/psychotropic medication for >=2 months and ongoing during treatment

Exclusion Criteria:

* Psychosis
* Bipolar I
* Acute suicidality
* Current substance use disorder
* Organic mental syndrome or intellectual disability
* Unstable non-HIV medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD Score based on the Clinician Administered PTSD Scale for DSM-5 | Baseline
  Lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS; diagnostic remission will be defined as achieving response plus failing to meet for DSM-5 defined PTSD per the CAPS after treatment.
Change in PTSD Score based on the Clinician Administered PTSD Scale for DSM-5 | Week 6
  Lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS; diagnostic remission will be defined as achieving response plus failing to meet for DSM-5 defined PTSD per the CAPS after treatment.
Change in PTSD Score based on the Clinician Administered PTSD Scale for DSM-5 | Week 12 (treatment termination)
  Lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS; diagnostic remission will be defined as achieving response plus failing to meet for DSM-5 defined PTSD per the CAPS after treatment.
Change in PTSD Score based on the Clinician Administered PTSD Scale for DSM-5 | 3-month post-treatment follow-up
  Lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS; diagnostic remission will be defined as achieving response plus failing to meet for DSM-5 defined PTSD per the CAPS after treatment.

SECONDARY OUTCOMES:
Change in Depression Score based on the Hamilton Depression Rating Scale (HDRS) | Baseline, Week 12 (treatment termination)
  The HDRS (also known as the Ham-D) scale contains 17 items pertaining to symptoms of depression experienced over the past week. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal, 8-16 suggest mild depression, 17-23 moderate depression, and scores over 24 are indicative of severe depression with the maximum score being 52 on the 17-point scale.
Change in Anxiety Score based on the Hamilton Rating Scale for Anxiety (HAM-A) | Baseline, Week 12 (treatment termination)
  Severity of anxiety will be assessed using the Hamilton Rating Scale for Anxiety (HAM-A). The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe anxiety.
Change in Functional Impairment based on the Sheehan Disability Scale (SDS) | Baseline, Week 6, Week 12 (treatment termination), 3-month post-treatment follow-up
  The Sheehan Disability Scale is a composite of three self-rated items designed to measure the extent to which three major domains in the patient's life are functionally impaired by psychiatric or medical symptoms. The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school (0-10 scoring range), social life (0-10 scoring range), and family life (0-10 scoring range). A composite range of 0-30 is possible. Scores of ≥5 on any of the 3 individual scales and overall higher totals scores are associated with significant functional impairment.

OTHER OUTCOMES:
Change in Drug and/or Alcohol Problems based on the Short Inventory of Problems-Alcohol and Drugs (SIP-AD) | Baseline, Week 6, Week 12 (treatment termination), 3-month post-treatment follow-up
  The Short Inventory of Problems Alcohol and Drugs is a fifteen item instrument used to assess the self-reported consequences of alcohol and substance abuse. The format establishes whether consequences ever happened to the respondents and the frequency of occurrence of the consequences. Possible responses are scored on a 4-point scale (0 = Never; 1 = Once or a few times; 2 = Once or twice a week; 3 = Daily or almost daily) based on occurrences over the prior 3-month period. A higher composite total is indicative of increasingly severe consequences.
Attrition from treatment by end of therapy duration | Up to Treatment Termination (Week 12)
  Attrition from treatment will be evaluated by the failure to complete experimental psychotherapy intervention defined as attending at least 16 out of 24 TFPP sessions within the 12-week period OR patient declaring intention to not attend any further TFPP sessions during the 12-week period. The specific session in which the patient dropped out will be recorded.
Change in AIDS Clinical Trials Group Adherence Questionnaire | Baseline, Week 6, Week 12 (treatment termination), 3-month post-treatment follow-up
  Gives a 3D day for day measure of AIDS drug compliance. Bigger number are better (taking more doses of medicine)
Number of patients with clinical PTSD response based on the Clinician Administered PTSD Scale for DSM-5 | Baseline, Week 6, Week 12 (treatment termination), 3-month post-treatment follow-up
  Lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS; diagnostic remission will be defined as achieving response plus failing to meet for DSM-5 defined PTSD per the CAPS after treatment.
Change in salivary cytokines | Baseline, Week 12 (treatment termination), 3-month post-treatment follow-up
  Multiple cytokines will be assessed: 14-Plex Luminex Panel of cytokines IL-1α, IL-1β, IL-6, IL-8, IL-17, TNF, IFN-g, MCP-1, MIP-3α, MIP-1α, MIP-1β, RANTES, GMCSF and CXCL9. Interpretation is joint, complicated, and determined within subject
Change in salivary cortisol | Baseline, Week 12 (treatment termination), 3-month post-treatment follow-up
  normal morning cortisol level depends on the lab but is around 0.094-1.551 µg/dL. Interpretations are made with-in person.
Change in HIV Viral Load | Baseline, Week 6, Week 12 (treatment termination)
  Larger numbers are indicative of greater viral load and are worse
Change in Complex PTSD symptoms based on an International Trauma Interview | Baseline, Week 6, Week 12 (treatment termination), 3-month post-treatment follow-up
  Additional instrument based off of the CAPS-5, assessing ICD-11 defined Complex PTSD symptoms; additionally meeting for Complex PTSD is defined by having at least one clinically significant symptom in each of the 3 symptom domains.
Change in symptom-specific reflective functioning | Baseline, Week 6, Week 12 (treatment termination)
  Lower scores indicate worse dysregulation, improvement denoted by higher numbers

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Milrod, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehn M, Milrod B, Chen CK. Clinical Case of Trauma-Focused Psychodynamic Psychotherapy for a Veteran With PTSD and Race-Based Trauma. Am J Psychother. 2024 Sep 1;77(3):146-150. doi: 10.1176/appi.psychotherapy.20230040. No abstract available. PMID 39277802